CLINICAL TRIAL: NCT01200095
Title: Non-hardware Posterior Cruciate Ligament Reconstruction Using Knot/Press-fit Technique With Periosteum-Evenloping Hamstrings Tendon Autograft
Brief Title: Posterior Cruciate Ligament Reconstruction Using Knot/Press-fit Technique
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Tai-Yuan Chuang, Department of Traumatology
Other Study IDs: 99045
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: PCL TEAR

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study presents an arthroscopic-assisted PCL reconstruction using femoral knot/press-fit technique with a periosteum-enveloping graft in tibial tunnel. The investigators evaluated the results of patients with PCL ruptures, who undergoing PCL reconstruction using this unique technique.

ELIGIBILITY:
Inclusion Criteria:

* PCL TEAR

Exclusion Criteria:

* PL INSTBILITY

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with PCL tear who received surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2003-01; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Yuan Chuang, Principal Investigator — Taipei Medical University WanFang Hospital